CLINICAL TRIAL: NCT03686748
Title: Retuning the Nervous System in Youth With Chronic Pain
Brief Title: Two Point Discrimination
Acronym: TPD
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Robert Coghill, Director of Research, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIN_TPD_001
Record Dates: First submitted 2018-06-27; First posted 2018-09-27 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Ehlers-Danlos Syndrome (EDS); Complex Regional Pain Syndrome (CRPS); Amplified Musculoskeletal Pain Syndrome (AMPS); Low Back Pain; Fibromyalgia; Chronic Widespread Pain
Keywords: Pain
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Complex Regional Pain Syndromes; Chronic Pain; Low Back Pain; Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: Two group, single blind for chronic pain patients receiving intervention, additional basic science component with baseline comparisons between patients and healthy controls.
Who Masked: Participant
Masking Description: Participant in the Chronic Pain Group are initially blinded to the intervention they will be receiving in the study.
  Healthy participants under go all assessments in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Two-point intervention (Experimental): Two point discrimination training.
  Interventions: Behavioral: Two-point discrimination training
- One-point intervention (Active Comparator): One point discrimination of size of probe
  Interventions: Behavioral: One-point discrimination training
- Healthy Controls (No Intervention): Observational component of differences in discrimination between chronic pain patients and healthy controls.

INTERVENTIONS:
Behavioral: Two-point discrimination training — Patients will undergo multiple sessions of two-point discrimination training.
  Arms: Two-point intervention
Behavioral: One-point discrimination training — Patients will undergo multiple sessions of one-point discrimination training.
  Arms: One-point intervention

SUMMARY:
SPECIFIC AIMS

Pain in both youth and adults is a complex, subjective and personal experience, and remains poorly understood. One particularly perplexing dimension of some forms of pain is the tendency of pain to spread outside of an affected body site to adjacent location, and then to unaffected body sites. Such widespread pain may reflect an altered spatial tuning of somatosensory processing, such that lateral inhibition is diminished, thereby allowing pain to spread. To date, no therapies exist which are designed specifically to diminish or even reverse the spatial spread of pain. However, training in two-point discrimination holds the potential to retune spatial aspects of somatosensory processing and may represent a novel therapy for widespread pain. Thus, the present investigation will test the following aims:

Aim 1. Do youth with chronic pain have disrupted spatial tuning of somatosensory processing? Deficits in two point tactile discrimination have long been noted in adults with chronic pain, but such deficits remain poorly documented in pediatric chronic pain patients. In order to determine if such deficits exist, youth with both chronic pain and healthy youth will undergo assessment of two point discrimination thresholds.

Aim 2. Does two-point discrimination training result in diminished pain and disability in youth with somatic pain? After initial characterization of tactile discrimination thresholds, youth with chronic pain will participate in multiple sessions of either two-point discrimination training or a single-point spatially-directed attentional control condition. Training will involve up to 9 additional sessions. Efficacy of training will be assessed by 1) reductions in the spatial extent of pain, 2) reductions in pain intensity and unpleasantness, and 3) reductions in pain-related disability.

DETAILED DESCRIPTION:
STUDY DESIGN Prior to commencing this investigation, investigators will optimize the tactile discrimination threshold testing (i.e. as per baseline visit, below), and the training conditions, in up to ten participants (patients and/or healthy controls). This will serve as a pilot to refine operational aspects of study procedures before investigators commence the main investigation proposed herein. Following this, youth with either chronic pain (ages 10-17, n=40) or healthy youth (ages 10-17, n=20) will undergo assessments of two-point and single-point discrimination thresholds in an initial session (Aim 1). After this initial session, youth with chronic pain will participate in up to 9 additional sessions of attentional training (Aim 2). These chronic pain patients will be randomized to either two-point discrimination training (n=20) or a single-point spatially-directed attentional control condition (n=20). Participants will not be informed of which intervention they will receive (single-blind study). Psychological questionnaires will be completed in the first and last sessions in order to determine how these variables relate to tactile discrimination and response to training.

STUDY INTERVENTIONS 5.1 Two Point Discrimination Training: Two-point discrimination threshold (TPD) training may be performed 1) at spatial locations remote from pain, 2) at spatial locations adjacent to the region of pain, and/or 3) at spatial locations in the site of pain, if the participant will tolerate it. TPD is defined as the smallest distance between two points at which someone can recognize two points, and not one, touching their skin. As such this is a test of one's ability to identify separate stimulation of two discrete areas, and relies heavily on lateral inhibition. Highly precise mechanical calipers will be gently placed onto the skin and the distance between the prongs will be increased/decreased. After repeated decreases and increases in the distance between the prongs, the TPD will be deemed as the distance at which participants consistently report two points instead of one. One-point stimuli will be interleaved to serve as a control condition. Participants will be informed immediately of correct and incorrect responses as part of the discrimination training.

5.2 Control Stimulation: Participants will undergo a single-point discrimination training at the same sites as described above. Probes of different sizes will be used for this portion - a small diameter probe (~1-5 mm) and a large diameter probe (~6-50mm). The probes will be gently placed in contact with the participants' skin, and the participant will be instructed to respond if they were contacted with the small or large probe. Participants will be informed immediately of correct and incorrect responses as part of the discrimination training.

ELIGIBILITY:
Inclusion Criteria:

Chronic Pain Patients:

* Somatically located chronic pain
* amplified musculoskeletal pain syndrome
* complex regional pain syndrome
* low back pain
* fibromyalgia
* other forms of chronic, widespread pain
* Male or female, 10-17 years
* High fluency in written and oral English language

Control Participants:

* Youth in good general health
* Male or female, 10-17 years
* High fluency in written and oral English language

Exclusion Criteria:

* Present significant mental health disorder as defined by DSM V (e.g. psychosis, bipolar disorder, major depression),
* alcohol or drug dependence
* documented developmental delays or impairments (e.g., autism, cerebral palsy, or mental retardation) of a magnitude that would interfere with adherence to study requirements or safe participation in the study
* Primary complaint of migraine or visceral (abdominal) pain, with minimal somatic involvement.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-07-21 (Actual); Primary Completion 2026-07-17 (Estimated); Study Completion 2027-07-16 (Estimated)

PRIMARY OUTCOMES:
Change in spatial extent of pain from baseline visit to final visit | baseline to final visit which is up to 5 weeks from baseline
  total area of body affected by pain
Change in pain ratings from baseline visit to final visit | baseline to final visit which is up to 5 weeks from baseline
  Ratings of current pain intensity on a non-numerical visual analog scale ranging from "not at all intense" to "most intense pain sensation imaginable" and of pain unpleasantness on a non-numerical visual analog scale ranging from "not at all unpleasant" to "most unpleasant pain imaginable".
Change in pain-related disability from baseline visit to final visit | baseline to final visit which is up to 5 weeks from baseline
  pain-related disability as assessed by the Functional Disability Index

SECONDARY OUTCOMES:
Change in two point discrimination threshold from baseline visit to final visit | baseline to final visit which is up to 5 weeks from baseline
  Calipers moving at fixed distances to determine threshold of two point detection

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Coghill, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected deidentified IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately after publication with no end date.
Access Criteria: Researchers who provide a methodologically sound proposal and who sign a data sharing agreement.

REFERENCES:
- [Background] Flor H, Nikolajsen L, Staehelin Jensen T. Phantom limb pain: a case of maladaptive CNS plasticity? Nat Rev Neurosci. 2006 Nov;7(11):873-81. doi: 10.1038/nrn1991. PMID 17053811
- [Background] Defrin R, Pope G, Davis KD. Interactions between spatial summation, 2-point discrimination and habituation of heat pain. Eur J Pain. 2008 Oct;12(7):900-9. doi: 10.1016/j.ejpain.2007.12.015. Epub 2008 Feb 14. PMID 18280188
- [Background] Flor H, Denke C, Schaefer M, Grusser S. Effect of sensory discrimination training on cortical reorganisation and phantom limb pain. Lancet. 2001 Jun 2;357(9270):1763-4. doi: 10.1016/S0140-6736(00)04890-X. PMID 11403816
- [Background] Gardner EP, Martin JH, Jessell TM, Kandel ER, Schwartz JH (2000) Principles of neural science. New York: McGraw-Hill.
- [Background] Groenewald CB, Essner BS, Wright D, Fesinmeyer MD, Palermo TM. The economic costs of chronic pain among a cohort of treatment-seeking adolescents in the United States. J Pain. 2014 Sep;15(9):925-33. doi: 10.1016/j.jpain.2014.06.002. Epub 2014 Jun 19. PMID 24953887
- [Background] Hechler T, Wager J, Zernikow B. Chronic pain treatment in children and adolescents: less is good, more is sometimes better. BMC Pediatr. 2014 Oct 13;14:262. doi: 10.1186/1471-2431-14-262. PMID 25308551
- [Background] Hestbaek L, Leboeuf-Yde C, Kyvik KO, Manniche C. The course of low back pain from adolescence to adulthood: eight-year follow-up of 9600 twins. Spine (Phila Pa 1976). 2006 Feb 15;31(4):468-72. doi: 10.1097/01.brs.0000199958.04073.d9. PMID 16481960
- [Background] Huguet A, Miro J. The severity of chronic pediatric pain: an epidemiological study. J Pain. 2008 Mar;9(3):226-36. doi: 10.1016/j.jpain.2007.10.015. Epub 2007 Dec 21. PMID 18088558
- [Background] King S, Chambers CT, Huguet A, MacNevin RC, McGrath PJ, Parker L, MacDonald AJ. The epidemiology of chronic pain in children and adolescents revisited: a systematic review. Pain. 2011 Dec;152(12):2729-2738. doi: 10.1016/j.pain.2011.07.016. PMID 22078064
- [Background] Lotze M, Moseley GL. Role of distorted body image in pain. Curr Rheumatol Rep. 2007 Dec;9(6):488-96. doi: 10.1007/s11926-007-0079-x. PMID 18177603
- [Background] Maihofner C, Handwerker HO, Neundorfer B, Birklein F. Patterns of cortical reorganization in complex regional pain syndrome. Neurology. 2003 Dec 23;61(12):1707-15. doi: 10.1212/01.wnl.0000098939.02752.8e. PMID 14694034
- [Background] Maihofner C, Handwerker HO, Neundorfer B, Birklein F. Cortical reorganization during recovery from complex regional pain syndrome. Neurology. 2004 Aug 24;63(4):693-701. doi: 10.1212/01.wnl.0000134661.46658.b0. PMID 15326245
- [Background] Moseley LG, Zalucki NM, Wiech K. Tactile discrimination, but not tactile stimulation alone, reduces chronic limb pain. Pain. 2008 Jul 31;137(3):600-608. doi: 10.1016/j.pain.2007.10.021. Epub 2007 Dec 3. PMID 18054437
- [Background] O'Sullivan PB, Beales DJ, Smith AJ, Straker LM. Low back pain in 17 year olds has substantial impact and represents an important public health disorder: a cross-sectional study. BMC Public Health. 2012 Feb 5;12:100. doi: 10.1186/1471-2458-12-100. PMID 22304903
- [Background] Price DD (1999) Psychological mechanisms of pain and analgesia, 0 Edition. Seattle: IASP Press.
- [Background] Price DD, McHaffie JG, Larson MA. Spatial summation of heat-induced pain: influence of stimulus area and spatial separation of stimuli on perceived pain sensation intensity and unpleasantness. J Neurophysiol. 1989 Dec;62(6):1270-9. doi: 10.1152/jn.1989.62.6.1270. PMID 2600624
- [Background] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411
- [Background] Quevedo AS, Coghill RC. Attentional modulation of spatial integration of pain: evidence for dynamic spatial tuning. J Neurosci. 2007 Oct 24;27(43):11635-40. doi: 10.1523/JNEUROSCI.3356-07.2007. PMID 17959806
- [Background] Quevedo AS, Morch CD, Andersen OK, Coghill RC. Lateral inhibition during nociceptive processing. Pain. 2017 Jun;158(6):1046-1052. doi: 10.1097/j.pain.0000000000000876. PMID 28195854
- [Background] Wand BM, Di Pietro F, George P, O'Connell NE. Tactile thresholds are preserved yet complex sensory function is impaired over the lumbar spine of chronic non-specific low back pain patients: a preliminary investigation. Physiotherapy. 2010 Dec;96(4):317-23. doi: 10.1016/j.physio.2010.02.005. PMID 21056167

DOCUMENTS (3):
  • Study Protocol (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03686748/Prot_003.pdf
  • Informed Consent Form: Healthy Control (2017-10-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03686748/ICF_000.pdf
  • Informed Consent Form: Patient Population (2017-10-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03686748/ICF_001.pdf